CLINICAL TRIAL: NCT01748006
Title: The Correlation Between Filling Pressure, Cardiac Output and Plasma Copeptin in Patients With Systolic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Finn Gustafsson (Other)
Responsible Party: Sponsor-Investigator, Finn Gustafsson, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-1-2012-019
Record Dates: First submitted 2012-08-15; First posted 2012-12-12 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine analyses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood and urine samples
  Interventions: Other: Standard of care therapy for severe decompensated heart failure

INTERVENTIONS:
Other: Standard of care therapy for severe decompensated heart failure

SUMMARY:
The relationship between the activation of the vasopressin system and central hemodynamics in heart failure (including right and left heart filling pressures and cardiac output) is not clear. The investigators intend to examine the correlation between levels of copeptin and vasopressin and the central hemodynamic system in patients with advanced (class III or IV) heart failure. The investigators also aim to examine the relationship of selected cardiac biomarkers in blood and urine with cardiac filling pressures and cardiac output in patients with decompensated heart failure.

The study population will consist of 30 patients admitted to the Department of Cardiology at Copenhagen University Hospital. Only patients for whom the attending cardiologist has already decided upon right heart catheterization for clinical/treatment reasons will be recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Left ventricular ejection fraction < 40 %
3. Diagnosed symptomatic heart failure treated with heart failure medications for at least 30 days.
4. Clinical indication for right heart catheterization for clinical/treatment reasons
5. NYHA-class III-IV
6. Relevant heart failure treatment as tolerated by the patient

Exclusion Criteria:

1. Absence of clinical/treatment indication of right heart catheterization
2. Syndrome of Inappropriate Secretion of ADH (SIADH)
3. Recent acute myocardial infarction within the last 30 days
4. Presence of infection or inflammatory disease
5. Malignant disease
6. Pregnancy
7. Subjects unwilling or unable to provide written consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 30 patients with heart failure admitted to the Department of Cardiology at the Copenhagen University Hospital, Rigshospitalet,Dennmark. Only patients who are already referred to right heart catheterization by the attending cardiologist will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The correlation between levels of plasma copeptin and vasopressin with left ventricular filling pressure and cardiac output | Day 1

SECONDARY OUTCOMES:
The correlation between levels of plasma copeptin and vasopressin with urine aquaporin-2 concentration | Day 1
The correlation between New York Heart Association (NYHA) class and levels of plasma copeptin and vasopressin | Day 1
The correlation between biomarkers levels and survival free of transplantation- and left ventricular assist device insertion | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Cardiology, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Balling L, Goetze JP, Jung MH, Rossing K, Boesgaard S, Gustafsson F. Copeptin levels and invasive hemodynamics in patients with advanced heart failure. Biomark Med. 2018 Aug;12(8):861-870. doi: 10.2217/bmm-2017-0439. Epub 2018 Jul 30. PMID 30058349